CLINICAL TRIAL: NCT06078813
Title: Spine SABR - Dose-escalated Stereotactic Ablative Body Radiotherapy (SABR) for Solid Tumour Spine Metastases
Acronym: Spine-SABR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 20-03
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor Spine Metastases
Keywords: Solid Tumor Spine Metastases; Dose-Escalated Stereotactic Ablative Body Radiotherapy

STUDY DESIGN:
Intervention Model Description: Treatment will consist of image guided dose escalated SABR using a simultaneous integrated boost (SIB) delivered in two fractions adhering to organ at risk dose-volume histogram constraints. There will be three dose levels delivered to the Planning Target Volume_1 (PTV_1) in each treatment arm as follows: 28 Gy (14 Gy per fraction), 30 Gy (15 Gy per fraction) and 32 Gy (16 Gy per fraction). A lower dose of 20 Gy (10 Gy per fraction) will be delivered to the PTV_2 which will be defined according to international consensus guidelines (Cox et al., 2012). The dose to PTV_2 will remain the same through all dose levels. All doses are prescribed to the target volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low baseline VCF risk (Experimental): All of:
  * No VCF
  * Predominantly sclerotic lesion (as determined by the Investigator based on MRI)
  * Normal spinal alignment
  * <50% vertebral body involvement
  Interventions: Radiation: Radiation: image guided dose escalated SABR using a simultaneous integrated boost (SIB)
- High baseline VCF risk (Experimental): Any of:
  * Pre-existing VCF
  * Predominantly lytic lesion (as determined by the Investigator based on MRI)
  * Spinal deformity
  * ≥50% vertebral body involvement
  Interventions: Radiation: Radiation: image guided dose escalated SABR using a simultaneous integrated boost (SIB)

INTERVENTIONS:
Radiation: Radiation: image guided dose escalated SABR using a simultaneous integrated boost (SIB) — Treatment will consist of image guided dose escalated SABR using a simultaneous integrated boost (SIB) delivered in two fractions adhering to organ at risk dose-volume histogram constraints. There will be three dose levels delivered to the Planning Target Volume_1 (PTV_1) in each treatment arm as follows: 28 Gy (14 Gy per fraction), 30 Gy (15 Gy per fraction) and 32 Gy (16 Gy per fraction). A lower dose of 20 Gy (10 Gy per fraction) will be delivered to the PTV_2 which will be defined according to international consensus guidelines (Cox et al., 2012). The dose to PTV_2 will remain the same through all dose levels. All doses are prescribed to the target volume.

SUMMARY:
This study will look at treatment for patients that have already been diagnosed with cancer, but develop a new tumor(s) in the spine. Patients who are not recommended for surgery are usually treated with 5-10 sessions of radiotherapy to manage symptoms. For patients with a longer life expectancy (>6 months), it is better to give a higher dose of treatment to potentially improve the duration of pain relief, cancer control and potentially survival. Higher doses of radiotherapy, however, may also cause worse toxicity and side effects. This study will look at delivering higher doses of radiation in 2 sessions rather than 5-10, using a more modern, targeted technique called image-guided Stereotactic Ablative Body Radiotherapy (SABR). This method requires special equipment and expertise compared to the traditional radiotherapy and this has limited availability in Ireland. This study aims to find out the highest dose that is safe to be given to patients and carefully examine the side effects. These results will help create national and international guidelines to benefit all cancer patients. Patients will be monitored closely during treatment and for 2 years afterwards. Patients have been involved in developing the treatment protocol and the patient information leaflet. Patients will also be asked to fill in quality of life (QOL) questionnaires at certain timepoints during the study. It is anticipated that this study will support the delivery of high quality SABR to all cancer patients in Ireland, resulting in potentially better quality of life, symptom and tumor control.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedures
2. ≥ 18 years of age
3. Life expectancy > 6 months
4. ECOG (Eastern Cooperative Oncology Group) performance status (PS) 0-2
5. Histological diagnosis of malignant primary disease (excluding haematologic, seminomatous or small cell subtype)
6. Diagnosis of oligometastatic disease (OMD) or oligoprogressive disease (OPD) defined as:

   1. OMD where there are 1 to 5 metastatic lesions, with a controlled primary tumor being optional, but where all metastatic sites must be safely treatable (can be synchronous or metachronous to primary tumor diagnosis) with curative intent OR
   2. OPD with 1 to 5 lesions progressing on a background of widespread but stable metastatic disease OR
   3. Systemic therapy-induced OMD where there are 1 to 5 persistent lesions after systemic therapy, all safely treatable with SABR
7. Single spinal level from C1 to L5 to be treated for the purpose of the study (co-existing lesion(s) on non-consecutive spinal level(s) may receive RT at Investigator discretion, if deemed unlikely to interfere with study treatment and assessment of outcomes).
8. Stable spine assessed by Spinal Instability Neoplastic Score (SINS) (SINS 0-6, or SINS 7-12 and not for surgical intervention).
9. Bilsky Grade 0-1a (i.e. minimal (epidural impingement, without deformation of thecal sac) or no epidural disease) as confirmed by Radiation Oncologist
10. Able to lie flat in the treatment position for radiotherapy for up to 60 minutes
11. Females of childbearing potential must not be pregnant or lactating, and must be prepared to take adequate contraception methods during treatment. Males whose female partners are of childbearing potential must be prepared to take adequate contraception methods during treatment. Examples of effective contraception methods are a condom or a diaphragm with spermicidal jelly, or oral, injectable or implanted birth control

Exclusion Criteria:

1. Previous radiotherapy or surgery to the proposed SABR treatment site which is likely to interfere with treatment or assessment of outcomes (for radiotherapy, this includes prior thoracic radiotherapy to the lung or oesophagus which would result in overlap of fields if a T spine lesion will be treated)
2. Patients with symptomatic spinal cord compression or cauda equina syndrome, resulting in bony compression or epidural compression of the spinal cord or cauda equine, respectively
3. Patients with syndromes or conditions associated with increased radiosensitivity
4. Patients with radiosensitive histologies, e.g. myeloma or lymphoma
5. Contraindication to MRI, e.g. MRI-incompatible personal pacemaker in situ
6. Patients with pre-existing osteoporotic fractures of the spine
7. Prior treatment with any radionuclide within 30 days prior to registration
8. Patients who have received chemotherapy within 1 week prior to administration of protocol RT or who are expected/planned to receive chemotherapy during RT or within 1 week after completing protocol RT
9. Uncontrolled intercurrent illness that is likely to interfere with treatment or assessment of outcomes, or psychiatric illness/social situations that would limit compliance with study requirements
10. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study, or if it is felt by the research / medical team that the patient may not be able to comply with the protocol and follow-up schedule due to psychological, familial, sociological or geographical conditions
11. Significant or progressive neurological deficit such that emergency surgery or radiation required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
The establishment of the MTD of 2-fraction spine SABR in patients with oligometastatic or oligoprogressive solid tumor metastases of the spine, by the number of patients experiencing DLTs within six months after treatment. | From start of treatment to 6 months post treatment
  DLT rate will be calculated as the proportion of evaluable patients (along with the 95% CI) experiencing a DLT, among the total evaluable patients.
  All evaluable patients will be used in the DLT analysis which will be performed after they have been potentially followed for the 6-months observation period. Patients not evaluable will be reported separately. For each such patient, the reason for exclusion, protocol treatment received, and toxicities reported during the first year will be listed.

SECONDARY OUTCOMES:
Estimate local progression-free survival at 1 and 2 years post-treatment, using Magnetic Resonance Imaging (MRI). | Up to 2 years post treatment
  Post treatment response and outcomes using MRI at 3, 6, 9, 12, 15, 18, and 24 months post-RT will be evaluated.
  The same patients used for DLT analysis will be used in these analyses. Radiation site (treated per study protocol) PFS (i.e. local PFS) at 1 year will be considered the key efficacy endpoint.
  Local progression is progression within the radiation site treated per study protocol, as identified on serial imaging. When local progression is suspected, two or three MRI scans 6-8 weeks apart are recommended per Investigator discretion (in line with international consortium (SPINO guidelines) (Thibault et al., 2015)).
  * Local control may be defined as the absence of progression within the radiation site treated per study protocol on serial imaging (MRI).
  * Any new or progressive tumor within the epidural space
  * Neurological deterioration attributable to pre-existing epidural disease with equivocal increased epidural disease dimensions on MRI
Estimate 6-month, 1-year and 2-year post-treatment overall survival rates. | Up to 2 years post treatment
  The Kaplan-Meier method will be used to estimate overall survival at each dose level. Cox proportional hazards regression will be used to characterise overall survival rate as a function of dose. Overall survival will be measured from the date of study registration until the date of death due to any cause or censoring.
Estimate the pain flare incidence 1 week post-treatment (i.e. 1 week after 2nd SABR fraction) using the Numeric Pain Rating Scale (NPRS) 0-10. | 1 week post treatment
  Pain score (including acute pain flare) at the radiation site treated per study protocol (assessed by numerical pain rating score, 0-10) (time frame: 1 week post treatment). [with secondary endpoint 4:] The changes in raw scores and percent change will be assessed over time using the Wilcoxon Signed rank test.
Pain score at radiation site (treated per study protocol) at 4 weeks, 3 months, 6 months, 1 year and 2 years post-treatment, using the NPRS. | Up to 2 years post-treatment
  Pain score (including acute pain flare) at the radiation site treated per study protocol (assessed by numerical pain rating score, 0-10) (time frame: 1 week post treatment). The changes in raw scores and percent change will be assessed over time using the Wilcoxon Signed rank test.
Acute toxicity profiles of ≥Grade 2 toxicities at 1- and 4-weeks post treatment, and at 3 months post-treatment using NCI CTCAE V5 | Up to 3 months post-treatment
  Counts and frequencies will be provided for the worst grade toxicity experienced by the patient. Acute toxicity profiles of ≥Grade 2 toxicities and their relatedness to study RT will be calculated, summarised and presented in tabular format with proportions, plus 95% confidence intervals where appropriate, at 1 and 4 weeks post treatment and at 3 months post-treatment using NCI CTCAE V5.
Late toxicity profiles of ≥Grade 2 toxicities and DLTs at 6, 9, 12, 15, 18 and 24 months post-treatment using NCI CTCAE V5. | Up to 2 years post-treatment
  Counts and frequencies will be provided for the worst grade toxicity experienced by the patient. Late toxicity profiles of ≥Grade 2 toxicities at 6, 9, 12, 15, 18 and 24 months post treatment completion, will be calculated, summarised and presented in tabular format with proportions, plus 95% confidence intervals where appropriate, using NCI CTCAE V5.
Estimates of time to onset of ≥ Grade 2 and ≥ Grade 3 acute toxicities. | Up to 3 months post-treatment
  Time-to-event analyses will be conducted for time to onset of the worst grade ≥2 and grade ≥3 acute toxicities separately. Kaplan-Meier curves will be presented and median point estimates (with 95% Cis) will be reported. Patients free of an event at the time of analysis will be censored at last available toxicity assessment. Time to toxicity will be measured from treatment start date. Patients alive and free of event at the time of analysis and patients lost to follow-up will be censored at the last available assessment.

OTHER OUTCOMES:
Estimate median time to onset of post-SABR ≥ Grade 2 VCF and rates of post-SABR ≥ Grade 2 VCF at 1 and 2 years. VCF is assessed via MRI. | Up to 2 years post-treatment
  Time-to-event analyses will be conducted for time to onset of ≥ Grade 2 VCF. Kaplan-Meier curves will be presented and median point estimates (with 95% Cis) will be reported. Patients free of an event at the time of analysis will be censored at last available assessment.
  Cox proportional hazards regression will be used to assess baseline demographic or clinical variables as risk factors for post-SABR VCF and to develop a nomogram to estimate risk of VCF for future studies.
Type of intervention (surgery or kyphoplasty) in the setting of post-SABR VCF at 1 and 2 years. | The type of intervention (surgery or kyphoplasty) in the setting of post-SABR VCF at 1 and 2 years will be described.
  Up to 2 years post-treatment
QoL outcomes at 6-months and 1-year post SABR (compared to baseline) using EORTC QLQ-BM22 (EORTC Quality of Life Questionnaire for Patients with Bone Metastases (22 questions)). | Up to 1 year post-treatment
  The mean and standard deviation (SD) of the overall and domain- and symptom-specific QoL outcomes at 6-months and 1-year post SABR (compared to baseline) using EORTC QLQ-BM22 scores at baseline and 6 months' post treatment will be reported. Scoring will be performed in accordance with the published guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Faul, MBBS, Principal Investigator — Cancer Trials Ireland/ St Luke's Radiation Oncology Network
Locations (3):
- Ireland (3):
  - Bon Secours/UPMC, Cork
  - St Luke's Radiation Oncology Network (SLRON) at Beaumont Hospital, Dublin
  - Beacon Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No